CLINICAL TRIAL: NCT06306469
Title: Changes in Microbiota and Biochemical Markers in Healthy Subjects Before and After Meditation Practices in a Controlled Environment
Brief Title: Changes in Microbiota in Healthy Subjects Before and After Meditation Practices in a Controlled Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pranic Healing Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PHRI-2022-1001
Record Dates: First submitted 2024-02-28; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Healthy
Keywords: microbiome; meditation; arhatic yoga; beneficial microbes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single Arm1 (Experimental): All practitioners had undertaken formal training on Pranic Healing, Meditation on Twin Hearts, and higher meditation practices at least six months prior to the retreat. Daily retreat practices, which lasted typically for 16-18 hours with occasional short breaks. These practices included combinations of specifically designed physical and breathing exercises to improve the energetic states and stillness. Exercises were followed by Pranic Healing and self-awareness practices. Meditations included Meditation on Twin Hearts, Arhatic Yoga meditations of Kundalini meditation, Arhatic Dhyan and Meditation on the Higher Soul .
  Interventions: Other: Meditation practice

INTERVENTIONS:
Other: Meditation practice — physical and breathing exercises

SUMMARY:
The goal of the study is to evaluate the Changes in Microbiota Markers in Healthy Subjects Before, During and After Meditation Practices in a Controlled Environment.

This study provides a unique opportunity to test the hypotheses that (1) Arhatic Yoga practices will affect both oral and gut microbiome; (2) the oral and gut microbiome will shift dynamically in a short period; and (3) the overall shift resulting from the changes in the gut microbiome members will be associated with known benefits to health and well-being.

DETAILED DESCRIPTION:
The present study was designed as a single-arm pilot scale to understand the temporal changes in both gut and oral microbiome of the practitioners at a meditation-cum-spiritual retreat in a controlled environment. There was open communication between all the participants before, during and after the retreat. As all the practitioners followed group practices in one location under the supervision of the senior instructors, separate assessment of the adherence of the practitioners to the protocol was not performed. Oral and fecal samples of practitioners were collected at the start (Day0: T1), middle (Day3-5: T2) and end (Day7-9:T3) of the retreat in a sterile containers. Amplicon sequencing was performed from extracted DNA to study changes in microbiome profile during retreat.

ELIGIBILITY:
Inclusion Criteria:

* must provide written informed consent prior to initiation of any study procedures
* was able to understand and agreed to comply with planned study procedures (agreed to the collection of specimens (saliva and fecal) before, during and after the study
* male or non-pregnant female greater than 18 years of age at time of enrolment
* must have a distinct Arhatic level (0-5 level) and performed meditation and MTH practices from once a week to more than 3 times a week prior to this retreat

Exclusion Criteria:

* concomitant disease that requires any medical treatment
* pregnancy
* any antibiotic treatment in the past two weeks
* pediatric population
* clinical apparent infectious disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-07-02 (Actual); Primary Completion 2022-07-09 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Assessing the changes in gut and oral microbiome profile of the participants during retreat | Timepoint1: 1 day (Baseline), Timepoint2: 3-5 days, and Timepoint3: 7-9 days
  Stool and oral samples were collected from the participants for three timepoints (T1: 1 day, T2: 3-5 days, and T3: 7-9 days) and changes in gut microbiome and oral microbiome were assessed through 16S rRNA gene amplicon sequencing. T1 was considered as baseline data.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Mendoza, Principal Investigator — Pranic Healing Research Institute,New Jersey, 07071, USA
Locations (1):
- Pranic Healing Research Institute, Lyndhurst, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Share the study protocol as well as raw data generated for amplicon sequencing
Supporting Information: Study Protocol, CSR
Time Frame: After publication, raw amplicon data will be available in NCBI for a very long time
Access Criteria: Bioproject ID from NCBI will be described in publication. Researchers can use that ID and download or see the data.

REFERENCES:
- [Background] Hammerschlag R, Sprengel ML, Baldwin AL. Biofield therapies: Guidelines for reporting clinical trials. Complement Ther Med. 2024 Jun;82:103011. doi: 10.1016/j.ctim.2023.103011. Epub 2024 Feb 1. PMID 38307809
- [Background] Raman M, Vishnubhotla R, Ramay HR, Goncalves MCB, Shin AS, Pawale D, Subramaniam B, Sadhasivam S. Isha yoga practices, vegan diet, and participation in Samyama meditation retreat: impact on the gut microbiome & metabolome - a non-randomized trial. BMC Complement Med Ther. 2023 Apr 5;23(1):107. doi: 10.1186/s12906-023-03935-8. PMID 37020274
- [Background] Househam AM, Peterson CT, Mills PJ, Chopra D. The Effects of Stress and Meditation on the Immune System, Human Microbiota, and Epigenetics. Adv Mind Body Med. 2017 Fall;31(4):10-25. PMID 29306937